CLINICAL TRIAL: NCT00893113
Title: A Phase 3, Double Blind, Placebo-Controlled, Crossover Study to Evaluate the Efficacy of Alfuzosin in Treating Men With ED and Mild LUTS.
Brief Title: An Efficacy Study to Evaluate Alfuzosin to Treat Men With Erectile Dysfunction and Mild Lower Urinary Tract Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chesapeake Urology Research Associates (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CURA-RT-002
Record Dates: First submitted 2009-04-08; First posted 2009-05-05 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Erectile Dysfunction; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Erectile Dysfunction; Lower Urinary Tract Symptoms | interventions — alfuzosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo, Then Alfuzosin (Placebo Comparator): Participants first received 1 Placebo tablet once daily for 12 weeks. Participants then received a 10 mg tablet of Alfuzosin daily for 12 weeks.
  Interventions: Drug: Placebo; Drug: Alfuzosin
- Alfuzosin, Then Placebo (Experimental): Participants first received a 10 mg tablet of Alfuzosin once daily for 12 weeks. Participants then received 1 Placebo tablet once daily for 12 weeks.
  Interventions: Drug: Placebo; Drug: Alfuzosin

INTERVENTIONS:
Drug: Placebo — Alfuzosin-matched One tablet once daily
Drug: Alfuzosin — 10 mg once daily

SUMMARY:
The purpose of this study is to assess the effect of Alfuzosin in treating Erectile Dysfunction in men with mild lower urinary tract symptoms based upon a change from baseline in erectile function (EF) domain of International Index of Erectile Function (IIEF).

DETAILED DESCRIPTION:
This protocol is a placebo-controlled, double-blind, crossover trial. Patients will be screened and then randomized to Group A or Group B at a 1:1 ratio to receive a placebo tablet once daily or Alfuzosin (10 mg) daily for 12 weeks. Patients will then crossover with the original placebo group receiving Alfuzosin for 12 weeks and the original Alfuzosin group receiving placebo. At every visit the patients will complete an IIEF and an AUA symptom index.

ELIGIBILITY:
Inclusion Criteria:

* Male, 30-69 years of age
* Has mild to moderate Erectile Dysfunction with a score < 25 on EF domain in IIEF
* AUA score of less than or equal to 14
* Negative urinalysis with no evidence of a Urinary Tract Infection

Exclusion Criteria:

* Blood pressure < 90/50 or > 170/110
* Neurological disorder (MS, SCI, CVA, Parkinson's disease, ALS)
* Diabetes Mellitus
* History of PSA > 10
* History of confirmed or suspected prostate cancer
* History of Moderate/Severe Hepatic Insufficiency defined as > 2X ULN
* On Alpha Blocker or PDE 5 inhibitor within 2 weeks of randomization
* Receive treatment with other investigational agents within 30 days prior to enrollment

Ages: 30 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald F Tutrone, MD, Principal Investigator — Chesapeake Urology Research Associates
Locations (3):
- United States (3):
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Glen Burnie, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Private Urology Practice, recruited patients from June 2009 through May 2012
Pre-assignment Details: Prior or current therapies of Alpha Blocker or PDE 5 inhibitor 2 weeks prior to randomization or investigational agents 30 days prior to randomization excluded them. 11 participants screen failed.
Groups:
- Placebo, Then Alfuzosin: Placebo: one tablet daily first, then 10 mg Alfuzosin daily
- Alfuzosin, Then Placebo: Alfuzosin: 10 mg once daily first, then one Placebo tablet daily
Period: Overall Study
Arm/Group | Placebo, Then Alfuzosin | Alfuzosin, Then Placebo
Started | 36 | 38
Completed | 23 | 22
Not Completed | 13 | 16
Not completed — Lost to Follow-up | 4 | 8
Not completed — Early Termination | 1 | 1
Not completed — Withdrew Consent | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Then Alfuzosin | Alfuzosin, Then Placebo | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 37 | 72
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 55 [36 to 69] | 53 [38 to 68] | 54 [36 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 36 | 38 | 74
Region of Enrollment [Number; unit: participants]
  United States | 36 | 38 | 74

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Erectile Function Domain of the International Index of Erectile Function
Description: The International Index of Erectile Function (IIEF) is used for the evaluation of male sexual function and diagnostic evaluation of Erectile Dysfunction (ED) severity. There are 5 domains of the IIEF: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. The Erectile Function (EF) domain of the IIEF is used to assess specific key components of ED including ability to achieve penetration and ability to maintain erection sufficient for satisfactory sexual performance. A score of 0-5 is awarded to each question of the IIEF. The EF domain pertains to questions 1, 2, 3, 4, 5, and 15. Scores are totaled and ranges are assigned to results. In the EF domain, a score of 0-30 is possible. The EF scores can be interpreted as follows: 0-6 severe dysfunction, 7-12 moderate dysfunction, 13-18 mild to moderate dysfunction, 19-24 mild dysfunction, and 25-30 no dysfunction.
Time Frame: Baseline and 12 Weeks
Population: The evaluable set includes all subjects who have sufficient data to assess the primary efficacy endpoint, and who have no major protocol deviations. Subjects were analyzed according to randomized treatment. Data for 45 subjects was analyzed.
Measure: Mean (Standard Deviation); unit: Change in EF Domain Score from Baseline
Groups:
- Placebo: Participants who received Placebo tablet (matching Alfuzosin 10 mg) in either the first or last 12 weeks of the study.
- Alfuzosin: Participants who received Alfuzosin 10 mg table in either the first or last 12 weeks of the study.
Arm/Group | Placebo | Alfuzosin
Number analyzed (Participants) | 23 | 22
Change in EF Domain Score from Baseline | 2.84 (7.492) | 2.84 (8.704)

2. Secondary Outcome: Changes in American Urological Association (AUA) Symptom Index
Description: The American Urological Association (AUA) Symptom Index is used to evaluate the severity of the patient's enlarged prostate symptoms. The AUA Symptom Index is completed by the patient. Questions are based on patient experiences in the past month and are answered on a scale of 0-5 (0 = not at all, 1 = less than one time in 5, 2 = less than half the time, 3 = about half the time, 4 = more than half the time, 5 = almost always). The scores are totaled and ranked as follows: mild (1-7), moderate (8-19), and severe (20-35).
Time Frame: Baseline and 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in AUA Score From Baseline
Arm/Group | Placebo | Alfuzosin
Number analyzed (Participants) | 23 | 22
Change in AUA Score From Baseline | -.1333 (4.984) | .4222 (5.345)

3. Secondary Outcome: Change in Total International Index of Erectile Function (IIEF) Score
Description: The International Index of Erectile Function (IIEF) is used for the evaluation of male sexual function and diagnostic evaluation of Erectile Dysfunction (ED) severity. There are 5 domains of the IIEF: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. A score of 0-5 is awarded to each question of the IIEF. Total IIEF scores range from 0-75. Lower scores indicate severe erectile dysfunction (0=severe erectile dysfunction), while higher scores indicate less erectile dysfunction (75=no erectile dysfunction).
Time Frame: Baseline and 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in Total IIEF Score from Baseline
Arm/Group | Placebo | Alfuzosin
Number analyzed (Participants) | 23 | 22
Change in Total IIEF Score from Baseline | 4.644 (14.872) | 6.24 (15.876)

ADVERSE EVENTS:
Time Frame: Every 12 weeks for each intervention.
Description: Adverse Events (AEs) were assessed at each visit by interviewing the patient. The Investigator assessed each AE and the relationship to the drug. AEs were only recorded if they were not listed on the label of Alfuzosin as a potential side effect.
Arm/Group | Placebo, Then Alfuzosin | Alfuzosin, Then Placebo
Serious Adverse Events (participants affected / at risk) | 1/36 | 1/38
Other Adverse Events (participants affected / at risk) | 0/36 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo, Then Alfuzosin (N=36) | Alfuzosin, Then Placebo (N=38)
Syncope (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — The assesment in the hospital revealed unclear etiology and the subject was discharged with a treatment plan to continue with pre admission medications, activity and diet. The subject was discontinued from the trial via withdrawal of consent
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient was admitted to the hospital for Shortness of Breath, pleuritic right sided chest pain. Patient was discontinued from trial via Investigator discretion.

LIMITATIONS AND CAVEATS:
Data compiled in this study is unable to neither prove nor disprove the objectives set. Placebo effect and recall bias may affect results. Regular sexual interaction and prior exposure to Alfuzosin were not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes